CLINICAL TRIAL: NCT07347977
Title: Lidocaine Infusion Decreases Postoperative Lung Cancer Reoccurance and Metatasis Risk: a Multicenter Randomized Controlled Study
Brief Title: Lidocaine Decreases Postoperative Lung Cancer Reoccurance and Metatasis Risk
Acronym: LidCRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, Changshun Huang, MD, Departmental director, First Affiliated Hospital of Ningbo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025B024
Record Dates: First submitted 2025-12-05; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Recurrence; Survival Analysis
Keywords: Lidocaine; Non-small cell lung cancer; Recurrence; Survival analysis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A random coding table is generated by statistical analysts, placed in a sealed and opaque envelope, and managed by an independent randomization specialist. The randomization specialist configures the medication according to the coding information, attaches the coding, and then provides it to the blinded anesthesiologist. Both patients, investigators and postoperative follow-up personnel are also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocine infusion group (Experimental): Lidocaine is administered intravenously at an ideal body weight (IBW) of 1.5 mg/kg starting from anesthesia induction, for 10-20 minutes, and then continuously infused at 1-1.5 mg/kg/h until 1 hour after skin closure, with a maximum rate of 120 mg/h. Use ideal weight instead of actual weight to prevent toxicity in very overweight patients. In patients with a weight lower than the ideal weight, the actual weight should be used to calculate the dose.
  Interventions: Drug: Lidocaine (drug)
- normal saline group (Placebo Comparator): The normal saline is administered at the volume calculated based on the equivalent volume of lidocaine dose according to body weight
  Interventions: Drug: Lidocaine (drug)

INTERVENTIONS:
Drug: Lidocaine (drug) — According to the random number table, grouping and coding are set, and the coding rules are predetermined by the statistical analyst. The intervention information is placed in a sealed opaque envelope and managed by an independent randomization specialist. After signing the informed consent form, the randomization specialist will configure drugs based on the grouping information and label them with codes, and hand them over to the anesthesiologist conducting blind intervention operations
  Other Names: Lidocaine IV

SUMMARY:
The goal of this clinical trial is to explore if perioperative lidocaine infusion decreases disease reoccurrence and metastasis risk in non-small cell lung cancer patients.

Participants will be randomly assigned (1:1) to the lidocaine or placebo group. The intervention initiates within 30 minutes before anesthesia induction with an intravenous loading dose of 1.5 mg/kg administered over 10-20 minutes. This is followed by a continuous maintenance infusion of 1.5-3 mg/kg/h (calculated as 1-1.5 mg/kg/h in protocol text, see note below) during surgery, terminating 1 hour after skin closure. Participants will be followed up for 36 months post-surgery. Blood samples will be collected at baseline, postoperative day 1, day 3, and upon discharge

DETAILED DESCRIPTION:
1. Research design: This is a 1:1 parallel, double-blind (participants, investigators, and outcomes assessors) randomized controlled trial. Intravenous lidocaine or saline will be assigned to patients with lung cancer undergoing minimally invasive (thoracoscopic or robotic) surgery.
2. Research Methods:

   2.1. Intervention: 2% lidocaine hydrochloride or placebo (0.9% sodium chloride).

   2.2. Dose planning: The intervention initiates within 30 minutes before anesthesia induction with an intravenous loading dose of 1.5 mg/kg (ideal body weight, IBW) administered over 10-20 minutes. This is followed by a continuous maintenance infusion of 1-1.5 mg/kg/h during surgery, terminating 1 hour after skin closure. The maximum infusion rate is capped at 120 mg/h. IBW is used to calculate dosage to prevent toxicity in overweight patients; however, for patients weighing less than their IBW, actual body weight is used. Patients in the placebo group receive the same volume and rate as the treatment group.

   Dose Guidelines Based on IBW (Broca Index): Males: height (cm) - 100; Females: height (cm) - 105.

   2.3. Dose adjustment: No dosage changes are permitted. If systemic local anesthetic toxicity is suspected, the infusion must be stopped immediately and not resumed. Supportive care and lipid emulsion therapy will be provided. If infusion is interrupted due to mechanical issues (e.g., pump malfunction), it may be restarted at the original rate.

   2.4. Additional care and procedures: To minimize confounding, general anesthesia will be maintained using a balanced technique. Postoperative care follows the unit's standard Enhanced Recovery After Surgery (ERAS) protocol. Concurrent continuous infusion of other local anesthetics (e.g., epidural or wound catheters) is prohibited during the IMP infusion period.

   2.5. Postoperative analgesia management: After surgery, all patients will receive intravenous patient-controlled analgesia (or continuous infusion) with sufentanil (2 µg/kg diluted to 100 ml) at a background rate of 2 ml/h.

   2.6. Sample size calculation: Based on a median recurrence-free survival (RFS) of 18 months in the control group and an expected extension to 24 months in the treatment group, the estimated Hazard Ratio (HR) is 0.75 (representing a 25% risk reduction). With a two-sided alpha of 0.05 and 90% power, 635 patients per group are required. Adjusting for a 10% dropout rate, the total sample size is set at 1400 patients (700 per group).

   2.7. Randomization: Participants will be randomly assigned (1:1) using a minimization algorithm. Stratification factors include age (<45, 45-65, 65-80 years), gender, trial center, and pathological type of lung cancer.
3. Efficacy evaluation criteria: The primary efficacy endpoint is Disease-Free Survival (DFS) within 36 months post-surgery. Chest CT scans will be performed at 6, 12, 18, 24, and 36 months to assess recurrence or metastasis. Additionally, the FACT-L questionnaire will be used to assess cancer-specific quality of life.
4. Adverse events: The lidocaine dose and duration in this study align with international consensus statements on safety. The infusion is limited to the intraoperative period and ends 1 hour post-skin closure, minimizing accumulation risks. Safety monitoring will be conducted throughout the infusion. In the event of toxicity, lipid emulsion (20%) is available for immediate rescue following AAGBI guidelines.
5. Quality control and quality assurance: SOPs will be strictly followed. Since the IMP infusion ends 1 hour after skin closure, monitoring will primarily occur in the operating room and PACU. Data will be recorded using EDC software. The investigators aim to collect outcome data for all randomized participants according to the intention-to-treat principle.
6. Statistical analysis: Data will be analyzed using SPSS 21 based on the intention-to-treat (ITT) principle.

   Primary Analysis: The primary outcome (DFS at 36 months) will be analyzed using a multivariate Cox regression model to estimate the Hazard Ratio (HR) between the lidocaine and placebo groups, adjusting for covariates.

   Covariates: Age, gender, comorbidities, ASA classification, cancer stage, and neoadjuvant therapies.

   Survival Analysis: Kaplan-Meier curves and Log-rank tests will be used to compare survival distributions.

   Missing Data: Missing data will be handled using multiple imputation to ensure robustness.
7. Ethics: The study adheres to the Declaration of Helsinki and local regulations. Ethics committee approval is required prior to initiation. Written informed consent will be obtained from all participants, ensuring they understand the risks and their right to withdraw. Privacy and data confidentiality will be strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years old.
2. Electively undergo minimally invasive (thoracoscopic or robotic) surgery for the treatment of lung cancer
3. Is willing and capable of providing consent.

Exclusion Criteria:

1. Palliative surgery without intention of cure.
2. Extensive comorbidities (ASA IV).
3. Patients with known or suspected allergy to lidocaine.
4. Patients who are currently pregnant or breastfeeding.
5. Patients who may experience adverse reactions due to accumulation of lidocaine during intravenous infusion, as stated in the Summary of Product Characteristics (SmPC) for lidocaine.
6. Currently, there is abnormal liver function, with ALT or AST levels exceeding the laboratory reference range by a factor of 2.
7. Currently, there is severe renal insufficiency (serum creatinine ≥451umol/L or glomerular filtration rate (calculated using the MDRD formula) <30ml/min).
8. Epilepsy.
9. Patients with cardiac conduction abnormalities, including second-degree or third-degree heart block without a pacemaker, left bundle branch block, sick sinus syndrome, and pre-excitation syndrome (confirmed by medical history and electrocardiogram), as well as those with low cardiac output due to reduced left ventricular ejection fraction.
10. Concurrent use with continuous infusion of other local anesthetic drugs (such as epidural).
11. Patients who use drugs that may cause reasons for exclusion, including Class I and Class III antiarrhythmic drugs (such as mexiletine and amiodarone), cimetidine, and antiviral drugs. Eligibility will be determined by local clinicians and verified by clinical trial doctors.
12. Patients with body weight <40kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 36 months after operation
  DFS is defined as the time from the date of surgery to the first documentation of disease recurrence (including local recurrence, regional lymph node metastasis, or distant metastasis) or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 36month after operation
  Overall survival is defined as the time from randomization to death from any cause
EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) | Baseline, Postoperative Day 1, Day 3, Discharge, and at 6, 12, 18, 24, 36 months post-surgery
  The EQ-5D-5L is used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  The EQ-5D-5L index score is calculated using population-based preference weights and typically ranges from less than 0 (health states worse than death) to 1 (full health), with higher scores indicating better health-related quality of life.In addition, the EQ Visual Analogue Scale (EQ-VAS) records the participant's self-rated health on a vertical scale ranging from 0 (worst imaginable health) to 100 (best imaginable health), with higher scores indicating better perceived health.
Cancer-specific quality of life measured using the Functional Assessment of Cancer Therapy - Lung (FACT-L) | Baseline, Postoperative Day 1, Day 3, Discharge, and at 6, 12, 18, 24, 36 months post-surgery
  The FACT-L is a validated instrument that includes the Functional Assessment of Cancer Therapy - General (FACT-G) and a lung cancer-specific subscale. The total FACT-L score ranges from 0 to 136, with higher scores indicating better cancer-specific quality of life.

OTHER OUTCOMES:
Total length of hospital stay | Up to 36 months
  Total length of hospital stay, including readmission, up to 36 months
Changes in Serum Biomarkers | Baseline, postoperative Day 1, postoperative Day 3, and at hospital discharge (assessed up to 5 days postoperatively).
  Changes in pro-inflammatory cytokine levels (e.g., interleukin-6 [IL-6], tumor necrosis factor-alpha [TNF-α], matrix metalloproteinase-9 [MMP-9], and matrix metalloproteinase-2 [MMP-2]) from baseline.
Incidence of Perioperative Adverse Events and Pain Scores | From the end of surgery up to hospital discharge (approximately 7-10 days)
  Assessment of perioperative complications including nausea, vomiting, and delirium, as well as pain intensity assessed using the Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating greater pain intensity.
Incidence of Cardiovascular Events | At 6 months and 12 months post-surgery
  Documentation of any new-onset cardiovascular events (e.g., arrhythmia, myocardial infarction) occurring after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Changshun Huang, MD, Principal Investigator — First Affiliated Hospital of Ningbo University
Locations (1):
- The first affiliated hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may not be shared because the informed consent does not include provisions for public data sharing, and data are subject to institutional and ethical review restrictions.

REFERENCES:
- [Result] Hiller JG, Perry NJ, Poulogiannis G, Riedel B, Sloan EK. Perioperative events influence cancer recurrence risk after surgery. Nat Rev Clin Oncol. 2018 Apr;15(4):205-218. doi: 10.1038/nrclinonc.2017.194. Epub 2017 Dec 28. PMID 29283170
- [Result] Ben-Eliyahu S, Golan T. Harnessing the Perioperative Period to Improve Long-term Cancer Outcomes. J Natl Cancer Inst. 2018 Oct 1;110(10):1137-1138. doi: 10.1093/jnci/djy055. No abstract available. PMID 29718287
- [Result] Wall TP, Buggy DJ. Perioperative Intravenous Lidocaine and Metastatic Cancer Recurrence - A Narrative Review. Front Oncol. 2021 Aug 2;11:688896. doi: 10.3389/fonc.2021.688896. eCollection 2021. PMID 34408981
- [Result] Zhang L, Hu R, Cheng Y, Wu X, Xi S, Sun Y, Jiang H. Lidocaine inhibits the proliferation of lung cancer by regulating the expression of GOLT1A. Cell Prolif. 2017 Oct;50(5):e12364. doi: 10.1111/cpr.12364. Epub 2017 Jul 24. PMID 28737263
- [Result] Chida K, Kanazawa H, Kinoshita H, Roy AM, Hakamada K, Takabe K. The role of lidocaine in cancer progression and patient survival. Pharmacol Ther. 2024 Jul;259:108654. doi: 10.1016/j.pharmthera.2024.108654. Epub 2024 May 1. PMID 38701900
- [Result] Manoleras AV, Sloan EK, Chang A. The sympathetic nervous system shapes the tumor microenvironment to impair chemotherapy response. Front Oncol. 2024 Sep 24;14:1460493. doi: 10.3389/fonc.2024.1460493. eCollection 2024. PMID 39381049
- [Result] Ramirez MF, Tran P, Cata JP. The effect of clinically therapeutic plasma concentrations of lidocaine on natural killer cell cytotoxicity. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):43-8. doi: 10.1097/AAP.0000000000000191. PMID 25469757
- [Result] Zhang H, Wang J, Li F. Modulation of natural killer cell exhaustion in the lungs: the key components from lung microenvironment and lung tumor microenvironment. Front Immunol. 2023 Nov 6;14:1286986. doi: 10.3389/fimmu.2023.1286986. eCollection 2023. PMID 38022613
- [Result] Piegeler T, Votta-Velis EG, Liu G, Place AT, Schwartz DE, Beck-Schimmer B, Minshall RD, Borgeat A. Antimetastatic potential of amide-linked local anesthetics: inhibition of lung adenocarcinoma cell migration and inflammatory Src signaling independent of sodium channel blockade. Anesthesiology. 2012 Sep;117(3):548-59. doi: 10.1097/ALN.0b013e3182661977. PMID 22846676
- [Result] Sullivan R, Alatise OI, Anderson BO, Audisio R, Autier P, Aggarwal A, Balch C, Brennan MF, Dare A, D'Cruz A, Eggermont AM, Fleming K, Gueye SM, Hagander L, Herrera CA, Holmer H, Ilbawi AM, Jarnheimer A, Ji JF, Kingham TP, Liberman J, Leather AJ, Meara JG, Mukhopadhyay S, Murthy SS, Omar S, Parham GP, Pramesh CS, Riviello R, Rodin D, Santini L, Shrikhande SV, Shrime M, Thomas R, Tsunoda AT, van de Velde C, Veronesi U, Vijaykumar DK, Watters D, Wang S, Wu YL, Zeiton M, Purushotham A. Global cancer surgery: delivering safe, affordable, and timely cancer surgery. Lancet Oncol. 2015 Sep;16(11):1193-224. doi: 10.1016/S1470-2045(15)00223-5. PMID 26427363
- [Result] Foo I, Macfarlane AJR, Srivastava D, Bhaskar A, Barker H, Knaggs R, Eipe N, Smith AF. The use of intravenous lidocaine for postoperative pain and recovery: international consensus statement on efficacy and safety. Anaesthesia. 2021 Feb;76(2):238-250. doi: 10.1111/anae.15270. Epub 2020 Nov 3. PMID 33141959
- [Result] Paterson H, Vadiveloo T, Innes K, Balfour A, Atter M, Stoddart A, Cotton S, Arnott R, Aucott L, Batham Z, Foo I, MacLennan G, Nimmo S, Speake D, Norrie J. Intravenous Lidocaine for Gut Function Recovery in Colonic Surgery: A Randomized Clinical Trial. JAMA. 2025 Jan 7;333(1):39-48. doi: 10.1001/jama.2024.23898. PMID 39602290

DOCUMENTS (2):
  • Study Protocol (2025-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT07347977/Prot_000.pdf
  • Informed Consent Form (2025-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT07347977/ICF_001.pdf